CLINICAL TRIAL: NCT03849950
Title: A Multi-Centre, Randomized Controlled Trial of Self-Management and Activation to Reduce Treatment-Related Toxicities in Patients Receiving Adjuvant or First-Line Metastatic Oral or Systematic Therapy for Colorectal, Lymphoma or Lung Cancer (SMARTCare)
Brief Title: Self-Management and Activation to Reduce Treatment-Related Toxicities (SMARTCare)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was halted prematurely due to the COVID-19 pandemic.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-SMARTCare-001
Record Dates: First submitted 2019-01-25; First posted 2019-02-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Lymphoma; Lung Cancer; Colo-rectal Cancer
Keywords: self-management support; health coaching; patient education; treatment-related toxicities
MeSH Terms: conditions — Lymphoma; Lung Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMARTCare (Experimental): 1. Training in self-management support (SMS) strategies for ambulatory nursing staff
  2. A web-based self-management education (I-Can-Manage Cancer) for patients
  3. Telephone-based, nurse-led health coaching
  4. Optional end of study patient interview (sub-study)
  Interventions: Other: SMARTCare
- Control (Active Comparator): 1. Training in self-management support (SMS) strategies for ambulatory nursing staff
  Interventions: Other: Control

INTERVENTIONS:
Other: SMARTCare — 1. Ambulatory nurses will undertake 4 hours of training consistent with the evidenced-based guidelines for SMS in routine care.
  2. An education program for patients in the intervention arm that targets training in core self-management skills and is comprised of an introduction and 5 education modules.
  3. An introductory call from a health coach prior to initiating treatment and 5 subsequent calls: prior to the first dose of treatment; 7-14 days following the first dose of treatment; within 2 weeks of coaching session 2; and timing is flexible for the last 2 sessions, but to be completed within 4 months following the first dose of treatment.
  4. Optional sub-study: A sub-set of patients will participate in an end of study interview to gain further insight into SMARTCare.
  Arms: SMARTCare
Other: Control — 1. Ambulatory nurses will undertake 4 hours of training consistent with the evidenced-based guidelines for SMS in routine care.
  Arms: Control

SUMMARY:
The investigators will undertake a multi-centre, randomized controlled trial to implement and evaluate a proactive model of care (SMARTCare) during active cancer treatment that incorporates self-management support (SMS). Patients allocated to the control arm will receive care from ambulatory clinic nurses trained in SMS. Patients allocated to the intervention arm will will receive care from ambulatory clinic nurses trained in SMS, in addition to being given access to a web-based, self-management education program and nurse-led health coaching during the first four months following the first systemic therapy administration.

DETAILED DESCRIPTION:
Self-management describes patient's behaviours and skills to manage the physical and psychosocial impact of their illness. Empirical evidence shows that patient activation in self-management results in improved disease control and quality of life (QOL), and lower emergency department visits and hospitalizations (ED+H) and costs in other chronic conditions. Previous research conducted by the investigators of this study has shown that the quality of SMS in ambulatory care was poor and patients felt unprepared to manage treatment-related toxicities. Building on previous work, this study will evaluate a multi-faceted proactive model of care that includes: (1) training in self-management support (SMS) strategies for ambulatory nursing staff; (2) a web-based self-management education program for patients; and (3) provision of proactive, nurse-led health coaching during the first four months following the first systemic therapy administration. Using a computer-generated permuted blocks randomization scheme (permuted blocks of random size) stratified by cancer type and centre, 160 evaluable patients will be enrolled across the three participating regional cancer centres. 80 patients will be randomized to the intervention arm and 80 to the control arm. The primary objective of this study is to compare the feasibility and acceptability of the SMARTCare intervention to the active comparator (control arm). The secondary objectives are to: (1) assess the effect of the intervention on symptom control, health-related quality of life, psychological distress, patient activation and self-efficacy; (2) evaluate the effect of the intervention on service outcomes: ED+H and resource utilization; and (3) evaluate implementation outcomes: fidelity, adherence and adoption. In addition, patients randomized to the intervention arm will be asked to participate in a sub-study interview at the end of the study to gain further knowledge about the SMARTCare intervention components from the patient's perspective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoma (Hodgkin's or non-Hodgkin's), colorectal, or lung cancer.
* Initiating adjuvant or first-line metastatic treatment with oral or systemic therapy within the accrual period at a participating centre. Patients receiving treatment with immunotherapy are eligible to participate.
* Eastern Cooperative Oncology Group (ECOG) </=2.
* Ability to understand and provide written informed consent.
* Access to an electronic device and internet connection to allow the participant to access the web-based I-Can-Manage Cancer education modules.
* Language and literacy skills consistent with completing validated questionnaires, and willingness to complete questionnaires as required.

Exclusion Criteria:

* Currently participating in a clinical trial involving receipt of an investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Reasons for non-participation | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Participating cancer centres will maintain Screening and Enrollment logs for the duration of the study. Reasons for non-participation will be documented on the logs and evaluated as one aspect of feasibility.
Reasons for premature discontinuation or withdrawal | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Reasons for premature discontinuation or withdrawal will be captured in MedidataRAVE and evaluated as one aspect of feasibility.
Recruitment rate | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Participating cancer centres will maintain Screening and Enrollment logs for the duration of the study. The logs will be used to calculate recruitment rates. The recruitment rate will be calculated as the proportion of patients that have agreed to participate among those approached and evaluated as one aspect of feasibility.
Retention rate | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Retention rate will be calculated as the proportion of patients who did not prematurely discontinue or withdraw among those that consented to participate, and evaluated as one aspect of feasibility.
Usage of I-Can-Manage (intervention arm only) | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Automated back-end analytics will be utilized to track patterns of usage of the I-Can-Manage Cancer Education Modules.
Compare the acceptability of the SMARTCare intervention to the active comparator by administering an Intervention Acceptability Questionnaire and conduct a thematic analysis of qualitative data from end of study interviews. | Assessed at 4-6 months post first dose +/- 2 weeks
  Acceptability of the intervention to patients will be evaluated using the Intervention Acceptability Questionnaire that has been developed for the study. The 3-section questionnaire (I-Can-Manage Cancer Modules; Health Coaching Calls; Overall Acceptability) asks patients to rate agreement statements from "Disagree Strongly" to "Agree Strongly". Individual scores for each statement in each section will be recorded.
  Audio recorded end of study qualitative interviews (approximately 30 minutes) will be conducted by a member of the study steering committee. The interviewer will follow a SMARTCare Patient Interview Guide. The guide consists of open-ended questions focusing on: (1) access, use, content and utility of the I-Can-Manage Cancer Modules; (2) logistics/timing/dose, content and utility of Health Coaching; and (3) General Comments. Interview transcripts will be analyzed in NVIVO to identify common themes.

SECONDARY OUTCOMES:
Patient Outcomes - Memorial Symptom Assessment Scale - Short Form (MSAS-SF) to evaluate the impact of the intervention on symptom control | Assessed at 2, 4 and 6 months post first dose +/- 2 weeks
  Patient outcomes will be evaluated using a series of questionnaires. To evaluate symptom control, the Memorial Symptom Assessment Scale - Short Form (MSAS-SF) will be administered. The MSAS-SF consists of a list of symptoms that patients answer "yes/no" to if they have experienced them in the past week. For symptoms answered yes, patients rate how much the symptom distressed or bothered them on a scale ranging from "Not at all (0)" to "Very Much (4)". The inclusion of this measure will allow the investigators and the study team to determine the best measure(s) to use as primary endpoint in the definitive trial.
Patient Outcomes - EQ-5D-5L to evaluate the impact of the intervention on health-related quality of life | Assessed at baseline and 2, 4 and 6 months post first dose +/- 2 weeks
  Patient outcomes will be evaluated using a series of questionnaires. To evaluate health-related quality of life, the EQ-5D-5L will be administered. The EQ-5D-5L consists of a series of headings with statements listed below. Patients are asked to select a box that best describes their health that day from a list of statements respective of each heading. The questionnaire also asks how good or bad their health is that day with 0 being the worst health a patient can imagine and 100 being the best health. The inclusion of this measure will allow the investigators and the study team to determine the best measure(s) to use as primary endpoint in the definitive trial.
Patient Outcomes - Hospital Anxiety and Depression Scale (HADS) to assess psychological distress | Assessed at baseline and 2, 4 and 6 months post first dose +/- 2 weeks
  Patient outcomes will be evaluated using a series of questionnaires. To evaluate psychological distress, the HADS will be administered. The HADS consists of different statements that patients are asked to respond to using a scale ranging from "Not at All (0)" to "Most of the time (3)". The inclusion of this measure will allow the investigators and the study team to determine the best measure(s) to use as primary endpoint in the definitive trial.
Patient Outcomes - Patient Activation Measure (PAM) to evaluate the impact of the intervention on patient activation | Assessed at baseline and 2, 4 and 6 months post first dose +/- 2 weeks
  Patient outcomes will be evaluated using a series of questionnaires. To evaluate patient activation, the PAM will be administered. The PAM consists of different statement that people sometimes make when they talk about their health. Patients are asked to respond to these statements using a scale ranging from "Disagree Strongly" to "Agree Strongly", or "N/A". The inclusion of this measure will allow the investigators and the study team to determine the best measure(s) to use as primary endpoint in the definitive trial.
Patient Outcomes - Patient Reported Outcomes Measurement Information System (PROMIS) short form to evaluate the impact of the intervention on self-efficacy | Assessed at baseline and 2, 4 and 6 months post first dose +/- 2 weeks
  Patient outcomes will be evaluated using a series of questionnaires. To evaluate self-efficacy, the PROMIS will be administered. The PROMIS consists of different self-efficacy confidence statements that patients are asked to respond to using a scale ranging from "I am not at all confident (1)" to "I am very confident (5)". The inclusion of this measure will allow the investigators and the study team to determine the best measure(s) to use as primary endpoint in the definitive trial.
System Outcomes - Impact of the intervention on incidence of emergency department visits and hospitalizations (ED+H) from administrative data. | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Emergency department visits and hospitalizations (ED+H) will be assessed using administrative data by linking patient-level data from the study to provincial administrative data using OHIP numbers.
  Information on drugs received, dates of treatment and institution where treatment was given will be identified from the Activity Level Reporting (ALR) database. The Ontario Cancer Registry (OCR) and the Collaborative Stage Database (CSD) will be used to confirm the patient has lymphoma, colorectal or lung cancer, as well as staging information. The National Ambulatory Care Reporting System (NACRS) database and Canadian Institutes for Health Information Discharge Abstract Database (CIHI-DAD) will be used to obtain information on ED visits and hospitalizations, respectively. All data analysis using healthcare administrative data will be completed at Cancer Care Ontario.
System Outcomes - Impact of the intervention on resource utilization (acute care visits and use of supportive care) from administrative data. | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Resource utilization will be compared between control and intervention arms using administrative data by linking patient-level data from the study to provincial administrative data using OHIP numbers.
  Information on drugs received, dates of treatment and institution where treatment was given will be identified from the Activity Level Reporting (ALR) database. The Ontario Cancer Registry (OCR) and the Collaborative Stage Database (CSD) will be used to confirm the patient has lymphoma, colorectal or lung cancer, as well as staging information. The National Ambulatory Care Reporting System (NACRS) database and Canadian Institutes for Health Information Discharge Abstract Database (CIHI-DAD) will be used to obtain information on ED visits and hospitalizations, respectively. All data analysis using healthcare administrative data will be completed at Cancer Care Ontario.
Implementation Outcomes - Fidelity of the intervention | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Members of the steering committee with expertise in health coaching will conduct two unannounced drop-in sessions at each of the participating centres to evaluate the content of the coaching calls, and health coaching reporting form documentation using a standardized evaluation form to take contemporaneous notes.
Implementation Outcomes - Patient adherence to the intervention | Assessed at baseline to 6 months post first dose +/- 2 weeks
  The proportion of calls delivered per protocol, based on information entered into MedidataRAVE will be calculated for each patient. Computerized back-end analytics will be used to capture how and when aspects of the I-Can-Manage Cancer Education Modules are accessed to evaluate patterns of usage.
Implementation Outcomes - Provider adoption of the intervention | Assessed at baseline to 6 months post first dose +/- 2 weeks
  Uptake of self-management support strategies will be analyzed using anonymous pre- and post-training evaluation form. Field notes will be used to track monthly meetings with participating cancer centres to summarize issues in implementation, and to inform mid-course correction to facilitate adoption of SMARTCare.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Krzyzanowska, MD MPH, Principal Investigator — University Health Network, Toronto; Doris Howell, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell D, Pond GR, Bryant-Lukosius D, Powis M, McGowan PT, Makuwaza T, Kukreti V, Rask S, Hack S, Krzyzanowska MK. Feasibility and Effectiveness of Self-Management Education and Coaching on Patient Activation for Managing Cancer Treatment Toxicities. J Natl Compr Canc Netw. 2023 Mar;21(3):247-256.e8. doi: 10.6004/jnccn.2022.7095. PMID 36898363